CLINICAL TRIAL: NCT06338709
Title: Clinical Study Protocol for the Assessment of Safety and Efficacy of the BARICLIP®
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Bariatric Technology (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-002
Record Dates: First submitted 2024-03-18; First posted 2024-04-01 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- BariClip® Device Treatment (Experimental): Subjects allocated to the Treatment Arm of this study will have a BariClip® device implanted.
  Interventions: Device: BariClip® Device Treatment
- Control (No Intervention): The implantation of a BariClip® device will not be performed on subjects allocated to the Control Arm of this study.

INTERVENTIONS:
Device: BariClip® Device Treatment — Device Administration (Implantation)
  Arms: BariClip® Device Treatment

SUMMARY:
Overweight and obesity are at epidemic proportions in the world population as well as in the United States, where nearly 42% of the adult population(1) is considered to meet the definition of obesity, namely a body mass index ("BMI") ≥ 30 kg/m2. Well-established links between obesity and increased morbidities and mortality make treatment of the utmost importance; however, there continues to be a significant unmet need for more effective treatments for obesity. Bariatric surgery is recognized as an effective treatment for obese patients, particularly in more severe cases where surgical restriction of the stomach's capacity and outlet size are considered necessary. The BariClip® is a laparoscopically implanted device for treatment of obesity and serves as an alternative to current existing technology for use in bariatric surgery. The BariClip® is a medical device, non-adjustable, resembling a clip that is placed parallel to the greater curvature of the stomach, causing restriction of the gastric lumen in a vertical fashion. This multi-center, randomized, moderate-lifestyle (program of diet and exercise) controlled pivotal study of the BariClip® device is intended to gather data to objectively support its safety and effectiveness for the treatment of obesity in adults and to ultimately support marketing authorization of this device as a viable alternative to existing bariatric surgical procedures. Specifically, this study aims to look at efficacy of the BariClip® device with regards to weight loss metrics and secondary health metrics and safety of the BariClip® device with regards to serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥22 years and ≤65 years
* Have signed an Informed Consent Form
* BMI 30-34.9 (with comorbidity) and 35-45 (with or without comorbidity) kg/m2
* Willing to comply with study requirements
* Subjects of childbearing potential not intending to become pregnant for the duration of their trial participation, with a documented negative pregnancy test and documentation of contraception confirmation and method
* History of obesity and being overweight (BMI >30kg/m2) for at least 1 year
* History of failure of non-surgical weight loss methods
* Fully ambulatory without any severe chronic orthopedic disease that requires reliance on crutches, walkers or a wheelchair that could preclude exercise during the study

Exclusion Criteria:

* Previous use of any device for the treatment of obesity
* Known hepatic disease or biliary disease prior to screening (e.g., viral, autoimmune, fibrosis /cirrhosis etiology, but not including incidental fatty liver)
* Known infection at time of randomization
* Enrolled in another investigational obesity study
* Uncorrectable bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet counts less than 100,000/microliter, or known coagulopathy
* Current substance abuse, alcohol or drug addiction
* Chronic pancreatitis or acute pancreatitis within 12 months of randomization
* Diagnosis of autoimmune connective tissue disorder (e.g., lupus erythematosus, scleroderma)
* Type I diabetes
* Hiatal hernia > 3cm
* Presence of ulcer in stomach
* Severe esophagitis (LA classification grade C or D)
* Presence of Barrett's esophagus
* Presence of any other abnormality that impacts the placement of the BariClip®
* Taking Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) (e.g., aspirin, ibuprofen, etc.) within 10 days prior to randomization and/or there is a need or expected need to use during the first 12 months after the index procedure
* Taking prescription antithrombotic therapy (e.g., anticoagulant, or antiplatelet agent) within 10 days prior to randomization and/or there is a need or expected need to use during the first 12 months after the index procedure
* Taking any of the medications on the list of Excluded Medications within 30 days prior to randomization and/or there is a need or expected need to use these medications during the first 12 months after the enrollment

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Achieving ≥ 5% total body weight loss (TBWL) in 50% of treated subjects | 12 months
Achieving ≥ 5% superiority margin for weight loss in the treated group as compared to the control group | 12 months

SECONDARY OUTCOMES:
Weight and Height will be combined to report BMI in kg/m^2 | 12 months
Blood Pressure (BP) in mmHg, both systolic and diastolic | 12 months
Diagnosis and/or Change in Severity of Diabetes Mellitus (DM) | 12 months
Weight in kilograms | 12 months
Height in meters | 12 months
Waist Circumference in centimeters | 12 months

OTHER OUTCOMES:
Incidence of Serious Adverse Events (SAEs) | Through study completion, total study duration estimated to be 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Moises Jacobs, MD, Study Director — Advanced Bariatric Technology

IPD SHARING:
Plan to Share IPD: Yes
To assess the safety and effectiveness of the Bariclip in patients with obesity.
Supporting Information: Study Protocol, CSR
Time Frame: Data available 1 year after last enrolled patient
Access Criteria: Access only to blinded study monitor until FDA approval of PMA